CLINICAL TRIAL: NCT01518998
Title: A Randomized, Double-Blind, Placebo-Controlled, 3x3 Factorial Design, Phase II Study to Evaluate the Antihypertensive Efficacy and Safety of Combination of Fimasartan and Amlodipine in Patients With Essential Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Collaborators: Gachon University Gil Medical Center (Other); The Catholic University of Korea (Other); Kyungpook National University Hospital (Other); Daegu Catholic University Medical Center (Other); Wonkwang University Hospital (Other); Wonju Severance Christian Hospital (Other); Korea University Guro Hospital (Other); DongGuk University (Other); Yeungnam University Hospital (Other); Chonnam National University Hospital (Other); Cheil General Hospital and Women's Healthcare Center (Other); Chungnam National University (Other); Asan Medical Center (Other); Seoul National University Bundang Hospital (Other); Inha University Hospital (Other); Seoul National University Hospital (Other); Inje University (Other); Samsung Medical Center (Other); Busan National University Yangsan Hospital (Unknown); Soon Chun Hyang University (Other); Catholic University of Korea Saint Paul's Hospital (Other); Hallym University Kangnam Sacred Heart Hospital (Other); Jeju National University Hospital (Other); Hanyang University Seoul Hospital (Other); Kangbuk Samsung Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: BR-FAC-CT-201
Record Dates: First submitted 2012-01-24; First posted 2012-01-26 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Hypertension
Keywords: Fimasartan; Amlodipine; antihypertension
MeSH Terms: conditions — Hypertension | interventions — fimasartan; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Placebo (Placebo Comparator): Take one double-blind capsule filled with a placebo tablet in the every morning
  Interventions: Drug: Fimasartan , Amlodipine, Placebo
- Fimasartan 60mg (Active Comparator): Take one double-blind capsule filled with of Fimasartan 60mg in the every morning
  Interventions: Drug: Fimasartan , Amlodipine, Placebo
- Fimasartan 30mg (Active Comparator): Take one double-blind capsule filled with Fimasartan 30mg in the every morning
  Interventions: Drug: Fimasartan , Amlodipine, Placebo
- Amlodipine 5mg (Active Comparator): Take one double-blind capsule filled with Amlodipine 5mg in the every morning
  Interventions: Drug: Fimasartan , Amlodipine, Placebo
- Amlodipine 10mg (Active Comparator): Take one double-blind capsule filled with Amlodipine 10mg in the every morning
  Interventions: Drug: Fimasartan , Amlodipine, Placebo
- Fimasartan 60mg/ Amlodipine 5mg (Experimental): Take one double-blind capsule filled with Fimasartan 60mg and Amlodipine 5mg in the every morning
  Interventions: Drug: Fimasartan , Amlodipine, Placebo
- Fimasartan 60mg/Amlodipine 10mg (Experimental): Take one double-blind capsule filled with Fimasartan 60mg and Amlodipine 10mg in the every morning
  Interventions: Drug: Fimasartan , Amlodipine, Placebo
- Fimasartan 30mg/Amlodipine 5mg (Experimental): Take one double-blind capsule filled with Fimasartan 30mg and Amlodipine 5mg in the every morning
  Interventions: Drug: Fimasartan , Amlodipine, Placebo
- Fimasartan 30mg/Amlodipine 10mg (Experimental): Take one double-blind capsule filled with Fimasartan 30mg and Amlodipine 10mg in the every morning
  Interventions: Drug: Fimasartan , Amlodipine, Placebo

INTERVENTIONS:
Drug: Fimasartan , Amlodipine, Placebo — Fimasartan 60mg, Fimasartan 30mg, Amlodipine 5mg, Amlodipine 10mg, Placebo, Fimasartan 60mg/Amlodipine 5mg combination, Fimasartan 60mg/Amlodipine 10mg combination, Fimasartan 30mg/Amlodipine 5mg combination, Fimasartan 30mg/Amlodipine 10mg combination
  Other Names: Kanarb; Norvasc

SUMMARY:
The purpose of this study is to evaluate the antihypertensive efficacy and safety of Fimasartan

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who agreed to participate in this study and submitted the written informed consent
2. Subjects aged 20 to 75 years
3. Essential hypertension subjects who are measured more 90mmHg, less than 114mmHg of sitting diastolic blood pressure (SiDBP) at baseline(day 0).
4. Subjects who considered to understand this study , be cooperative, and able to be followed-up whole of the study period.

Exclusion Criteria:

1. Severe hypertension patients; more 115mmHg of SiDBP and/or more 185 mmHg of Sitting systolic blood pressure (SiSBP)
2. Patients with secondary hypertension
3. Patients with significant investigations - abnormal renal function (Creatinine more 1.5 times than upper limit of normal), abnormal liver function (AST, ALT more 2 times than upper normal), moderate fatty lever needed medication
4. Patients with significant investigations - Hypokalemia(Less than 3.5mmol/L), Hyperkalemia(exceeded 5.5mmol/L)
5. Patients with sodium ion or body fluid is depleted and not able to correct
6. Patients with hypotension who has sign and symptom
7. Patients with surgical and medical disease it is able to be affect to absorption, distribution, metabolism, excretion
8. Patients with severe insulin dependent or uncontrolled diabetes mellitus (HbA1c > 9%, regimen change of oral hypoglycemic agent, using insulin)
9. Patients with severe heart disease, ischemic heart disease within 6months, peripheral vascular disease, Percutaneous Transluminal Coronary Angiography (PTCA), Coronary Artery Bypass Graft (CABG)
10. Patients with significant ventricular tachycardia, atrial fibrillation, atrial flutter or other significant arrhythmia
11. Patients with hypertrophic obstructive cardiomyopathy, severe obstructive coronary artery disease, aortic stenosis, hemodynamically significant aortic valve or mitral valve disease
12. Patients with severe cerebrovascular disease
13. Patients with wasting disease, autoimmune disease, connective tissue disease at present and/or previous.
14. Patients with known severe or malignancy retinopathy
15. Patients with hepatitis B or C or HIV positive reaction
16. Patients who have a story or evidence of alcohol or drug abuse within 2years
17. Patients who are measured the mean difference of mean blood pressure of both arm under SiDBP 10mmHg or SiSBP 20mmHg at screening and baseline visit
18. Patients with history of allergic reaction to any angiotensin II antagonist
19. Patients with any chronic inflammation disease needed to chronic inflammation therapy
20. Patients with the medical histories of malignant tumor within 5years, except local basal cell carcinoma of the skin
21. Childbearing and breast-feeding women
22. Female who plan to become pregnancy or have a possibility of pregnancy but don't prevent conception with acknowledged methods
23. Patients who took medicine within 12 weeks from screening visit or is going on the progress of other clinical trial
24. Subject who are judged unsuitable to participate in this study by investigator

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2011-08; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Sitting Diastolic Blood Pressure | 8weeks from baseline visit
  To compare the difference of Sitting Diastolic Blood Pressure at 8 weeks from baseline visit

SECONDARY OUTCOMES:
Sitting Systolic Blood Pressure | at 4 and 8 weeks from Baseline visit
  To compare the difference of Sitting Systolic Blood Pressure at 4,8 weeks from baseline visit
Sitting Diastolic Blood Pressure | 4weeks from baseline visit
  To compare the difference of Sitting Diastolic Blood Pressure at 4 weeks from baseline visit
Responder ratio | at 8weeks from baseline visit
  To compare the ratio or responder(SiDBP<90mmHg or difference of SiDBP>10mmHg from baseline) at 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Young Kwan Jeon, Medical Director, Study Director — Boryung Pharmaceutical Co., Ltd
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Lee HY, Kim YJ, Ahn T, Youn HJ, Chull Chae S, Seog Seo H, Kim KS, Rhee MY, Choi DJ, Kim JJ, Chun KJ, Yoo BS, Park JS, Oh SK, Kim DS, Kwan J, Ahn Y, Bae Park J, Jeong JO, Hyon MS, Cho EJ, Han KR, Kim DI, Joo SJ, Shin JH, Sung KC, Jeon ES. A Randomized, Multicenter, Double-blind, Placebo-controlled, 3 x 3 Factorial Design, Phase II Study to Evaluate the Efficacy and Safety of the Combination of Fimasartan/Amlodipine in Patients With Essential Hypertension. Clin Ther. 2015 Nov 1;37(11):2581-2596.e3. doi: 10.1016/j.clinthera.2015.02.019. Epub 2015 Apr 4. PMID 25850881